CLINICAL TRIAL: NCT06490484
Title: Efficacy and Safety of HSK16149 Capsule in Chinese Patients With Diabetic Peripheral Neuropathic Pain Who Had an Inadequate Response to Pregabalin: A Prospective, Multicenter, Randomized, Double-Blind, Double-Dummy, Pregabalin-controlled Phase 2 Study
Brief Title: Efficacy and Safety of HSK16149 Capsule in Chinese Patients With Diabetic Peripheral Neuropathic Pain Who Had an Inadequate Response to Pregabalin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK16149-207
Record Dates: First submitted 2024-06-10; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — BID protein, human; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK16149 20mg BID (Experimental): Drug: HSK16149 20mg BID HSK16149 20mg, orally twice a day; treatment period: 4 weeks fixed dose.
  Interventions: Drug: HSK16149 20mg BID
- Pregabalin 150 BID (Experimental): Drug: Pregabalin 150mg BID Pregabalin 150mg, orally twice a day; treatment period: 1 week titration and 3 weeks fixed dose.
  Interventions: Drug: Pregabalin 150mg BID

INTERVENTIONS:
Drug: HSK16149 20mg BID — Drug: HSK16149 20mg BID HSK16149 20mg, orally twice a day; treatment period: 4 weeks fixed dose.
  Other Names: Crisugabalin
  Arms: HSK16149 20mg BID
Drug: Pregabalin 150mg BID — Drug: Pregabalin 150mg BID Pregabalin 150mg, orally twice a day; treatment period: 1 week titration and 3 weeks fixed dose.
  Other Names: Pregabalin
  Arms: Pregabalin 150 BID

SUMMARY:
Investigate the efficacy and safety of HSK16149 capsule in Chinese patients with Diabetic Peripheral Neuropathic Pain (DPNP) who had an inadequate response to Pregabalin, following 4 weeks treatment in comparison to Pregabalin

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. Males or females aged 18-75 years of age inclusive;
3. Diagnosis of diabetic peripheral neuropathic pain (DPNP) and diabetic peripheral neuropathy (DPN) pain ≥ 6 months;
4. HbA1c ≤ 11.0% at screening and on a stable anti-diabetic medication regimen for at least 30 days prior to screening;
5. Have a visual analog scale (VAS) pain value ≥60 mm in the past 24 h during screening;
6. DPNP patients are currently receiving continuous treatment with pregabalin for more than 4 weeks who had an inadequate response.

Exclusion Criteria:

1. Peripheral neuropathy or pain unrelated to DPN that may confuse the assessment of DPNP.
2. Skin conditions in the area affected by neurupathy that could alter sensation.
3. Chronic systemic diseases that may affect subjects' participation in the study.
4. Severe hematologic, hepatic or renal dysfunction, the subject will be excluded if:

   1. Neutrophils < 1.5 × 10^9/L, or platelet < 90 × 10^9/L, or hemoglobin < 100 g/L;
   2. AST/ALT > 2.5 × upper limit of normal (ULN), or TBIL > 1.5 × ULN;
   3. Estimation of glomerular filtration rate (eGFR) < 60 mL/min / 1.73 m^2;
   4. Creatine kinase > 2.0 × ULN.
5. History of substance abuse or alcohol abuse.
6. Acute complications of diabetes in the 6 months prior to screening.
7. Any active infections at screening.
8. HBsAg or HCV Ab positive, or HIV Ab positive, or serum TP Ab positive.
9. Inability or unwillingness to discontinue any other prohibited concomitant medications.
10. History of allergic or medically significant adverse reaction to investigational products or their excipients, duloxetine or related compounds.
11. History of suicidal behavior or attempted suicide.
12. Pregnant or preparing for pregnancy or breastfeeding during the study period, or subjects were not willing to use reliable contraceptives methods from the date of ICF signature until 28 days after the last trial drug administration, or planning to use progesterone contraceptives during this period.
13. Participated in another clinical study within 30 days prior to screening.
14. Other conditions of the subjects who are unlikely to comply with the protocol.
15. The investigators determine that there are other conditions that are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-07-12 (Estimated); Study Completion 2024-07-14 (Estimated)

PRIMARY OUTCOMES:
Compare the change from baseline in Visual Analog Scale (VAS) between HSK16149 and Pregabalin at week 4. | Baseline and week 4
  The VAS, in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain.

SECONDARY OUTCOMES:
Compare the change from baseline in Numeric Rating Scales (NRS) between HSK16149 and Pregabalin at week 4. | Baseline and week 4
  The NRS, in which the participant rates pain on a 11-point numeric rating scale, where 0 = no pain and 10 = worst possible pain.
Compare the change from baseline in Visual Analog Scale (VAS) between HSK16149 and Pregabalin at treatment period. | Baseline to week 4
  The VAS, in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain.
Compare the change from baseline in Short-Form McGill Pain Questionnaire (SF-MPQ) betwwen HSK16149 and Pregabalin at week 4. | Baseline and week 4
  Participants rate their pain in three parts of the questionnaire, which are combined into a single pain intensity score:
  Part 1 - fifteen descriptors of pain intensity, on a scale of 0 (none) to 3 (severe);
  Part 2 - the VAS, in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain;
  Part 3 - a present pain intensity index in which the participant rates present pain intensity on a scale of 0 (no pain) to 5 (most intense pain).
Compare the change from baseline in Daily Sleep Interference Score (DSIS) between HSK16149 and Pregabalin at week 4. | Baseline and week 4
  The sleep interference scores on a scale of 0-10, where 0 = pain did not interfere with sleep to 10 = pain completely interfered with sleep. The weekly DSIS is based on participants daily sleep interference scores.
Compare the change from baseline in EuroQol-5-Domain-5-Level health questionnaire (EQ-5D-5L) between HSK16149 and Pregabalin at week 4. | Baseline and week 4
  The EQ-5D-5L assessed quality of life based on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant was asked to 'check the ONE box that best describes your health TODAY,' choosing from 5 options (no problems, slight problems, moderate problems, severe problems, extreme problems) provided under each dimension. The health state index value is a single value on a scale from 0 to 100 scores indicating better health: 0 = indicating worst health and 100 = best imaginable health.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No